CLINICAL TRIAL: NCT00407966
Title: Phase II Study of Alvocidib (NSC 649890, Flavopiridol) in Timed Sequential Combination With Cytosine Arabinoside (Ara-C) and Mitoxantrone for Adults With Newly Diagnosed, Previously Untreated, Poor-Risk Acute Myelogenous Leukemias
Brief Title: Alvocidib, Cytarabine, and Mitoxantrone in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02986; NCI-2012-02986 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U01CA070095 (NIH); P30CA006973 (NIH); J0669 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 7845 (Other: CTEP)
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2012-12

CONDITIONS: Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — alvocidib; Cytarabine; Mitoxantrone

ARMS (1):
- Treatment (alvocidib, cytarabine, mitoxantrone hydrochloride) (Experimental): Patients receive alvocidib IV over 1 hour on days 1-3, cytarabine IV continuously over 72 hours on days 6-8, and mitoxantrone hydrochloride IV over 1-2 hours on day 9. Beginning 35-63 days after completion of course 1, patients achieving complete or partial remission may receive a second course of treatment as above.
  Patients age 50 and over with "core binding factor" acute myeloid leukemia (AML) (e.g., t[8;21], inv[16], or t[16;16]) achieving a complete remission after course 1 of treatment may receive 3-4 courses of consolidation therapy comprising high-dose cytarabine at the discretion of the investigator.
  Interventions: Drug: alvocidib; Drug: cytarabine; Drug: mitoxantrone hydrochloride

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Novantrone

SUMMARY:
This phase II trial is studying the side effects and how well giving alvocidib together with cytarabine and mitoxantrone works in treating patients with newly diagnosed acute myeloid leukemia. Drugs used in chemotherapy, such as alvocidib, cytarabine, and mitoxantrone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy and toxicities of flavopiridol (alvocidib) followed by ara-C and mitoxantrone in adults with newly diagnosed acute myelogenous leukemia (AML) with poor-risk features.

II. To determine the disease free and overall survival of patients exhibiting a response to treatment with flavopiridol followed by ara-C and mitoxantrone.

OUTLINE:

Patients receive alvocidib IV over 1 hour on days 1-3, cytarabine IV continuously over 72 hours on days 6-8, and mitoxantrone hydrochloride IV over 1-2 hours on day 9. Beginning 35-63 days after completion of course 1, patients achieving complete or partial remission may receive a second course of treatment as above.

Patients age 50 and over with "core binding factor" acute myeloid leukemia (AML) (e.g., t[8;21], inv[16], or t[16;16]) achieving a complete remission after course 1 of treatment may receive 3-4 courses of consolidation therapy comprising high-dose cytarabine at the discretion of the investigator.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Adults with established, pathologically confirmed diagnoses of newly diagnosed, poor-risk Acute Myeloid Leukemia(AML) including de novo and secondary Acute Myeloid Leukemias but excluding newly diagnosed acute progranulocytic leukemia (APL, M3) will be considered eligible for study
* ECOG performance status 0-2
* Patient must be able to give informed consent
* Serum creatinine =< 2.0
* ALT, AST =< 5 x upper limit of normal
* Bilirubin =< 2.0 mg/dl
* Left ventricular ejection fraction >= 45%
* Newly diagnosed AML, subtypes M0,1,2,4-7 but excluding M3 (APL) with poor-risk features, including:

  * Age > 50 years, or age > 18 years with one or more of the following criteria:

    * Antecedent hematologic disorder including myelodysplasia (MDS)-related AML (MDS/AML) and prior myeloproliferative disorder (MPD)
    * Treatment-related AML
    * AML with trilineage dysplasia (AML-TLD)
    * Adverse cytogenetics (defined as -5/-5q; -7/-7q; abnormal 3q, 9q, 11q, 20q, 21q or 17p; t(6;9); t(9;22); trisomy 8; trisomy 13, complex karyotypes (>= 3 unrelated abnormalities)

Exclusion Criteria:

* Patients who have received hydroxyurea alone or have received non-cytotoxic therapies previously for MDS or MPD (e.g., thalidomide or lenalidomide, interferon, cytokines, low-dose 5-azacytidine, low-dose cytoxan) will be eligible for this trial
* Any previous treatment with flavopiridol
* Concomitant chemotherapy, radiation therapy, or immunotherapy
* Hyperleukocytosis with >= 50,000 blasts/uL; leukapheresis or hydroxyurea may be used immediately prior to study drug administration for cytoreduction; must be stopped 24 hours before first dose of Flavopiridol
* Acute Progranulocytic Leukemia (APL, M3)
* Active CNS leukemia
* Active, uncontrolled infection; patients with infection under active treatment and controlled with antibiotics are eligible
* Presence of other life-threatening illness
* Patients with mental deficits and/or psychiatric history that preclude them form giving informed consent or from following protocol
* Pregnant and nursing patients are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-10; Primary Completion 2008-07 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Karp, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (1):
- Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Karp JE, Garrett-Mayer E, Estey EH, Rudek MA, Smith BD, Greer JM, Drye DM, Mackey K, Dorcy KS, Gore SD, Levis MJ, McDevitt MA, Carraway HE, Pratz KW, Gladstone DE, Showel MM, Othus M, Doyle LA, Wright JJ, Pagel JM. Randomized phase II study of two schedules of flavopiridol given as timed sequential therapy with cytosine arabinoside and mitoxantrone for adults with newly diagnosed, poor-risk acute myelogenous leukemia. Haematologica. 2012 Nov;97(11):1736-42. doi: 10.3324/haematol.2012.062539. Epub 2012 Jun 24. PMID 22733022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 2006 through June 2008
Groups:
- Arm A: Flavopiridol, ara-C, mitoxantrone
Period: Overall Study
Arm/Group | Arm A
Started | 45
CR | 30
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm A
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Complete Response
Description: Bone marrow showing less than 5% myeloblasts with normal maturation of all cell lines, an Absolute Neutrophil Count of at least 1000/mililiter and a platelet count of 100,000 mililiter, absence of blast in peripheral blood, absence of identifiable leukemic cells in the bone marrow, clearance of disease-associated cytogenetic abnormalities, and clearance of any previously existing extramedullary disease. A complete remission must be confirmed 4 to 6 weeks after the initial documentation. If possible, at least one bone marrow biopsy should be performed to confirm the complete remission.
Time Frame: 6 months
Population: Total number of participants entered between December 2006 and June 2008
Measure: Number; unit: participants
Arm/Group | Arm A
Number analyzed (Participants) | 45
participants | 45

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of treatmetn through recovery of blood counts and response assessment
Arm/Group | Arm A
Serious Adverse Events (participants affected / at risk) | 19/45
Other Adverse Events (participants affected / at risk) | 25/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=45)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 19 (19)
cardiac dysfunction (Cardiac disorders) | 7 (7)
Desseminated Intravascular Coagulopathy (Investigations) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=45)
oral mucositis (Gastrointestinal disorders) | 14 (14)
Diarrhea (Gastrointestinal disorders) | 11 (11)
GI Mucositis (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less